CLINICAL TRIAL: NCT02140489
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate a Pharmacokinetic Drug Interaction Between Amlodipine/Losartan and Rosuvastatin in Healthy Male Volunteers
Brief Title: Evaluating a Pharmacokinetic Drug Interaction Between Amlodipine/Losartan and Rosuvastatin
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ALRO-101
Record Dates: First submitted 2014-03-09; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1 (Experimental): amosartan → rosuvastatin → amosartan and rosuvastatin
  Interventions: Drug: amosartan; Drug: rosuvastatin; Drug: amosartan and rosuvastatin
- Sequence 2 (Experimental): rosuvastatin → amosartan and rosuvastatin → amosartan
  Interventions: Drug: amosartan; Drug: rosuvastatin; Drug: amosartan and rosuvastatin
- Sequence 3 (Experimental): amosartan and rosuvastatin → amosartan → rosuvastatin
  Interventions: Drug: amosartan; Drug: rosuvastatin; Drug: amosartan and rosuvastatin

INTERVENTIONS:
Drug: amosartan
  Other Names: amosartan, P.O
Drug: rosuvastatin
  Other Names: rosuvastatin, P.O
Drug: amosartan and rosuvastatin
  Other Names: amosartan and rosuvastatin, P.O

SUMMARY:
The purpose of this study is to evaluate the drug-drug interaction between amlodipine/losartan and rosuvastatin in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Age between 19 and 55
* Signed informed consent

Exclusion Criteria:

* Presence of medical history or a concurrent disease
* Has a history of hypersensitivity to IP ingredients

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-05 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Cmax | 0-72h
AUClast | 0-72h

SECONDARY OUTCOMES:
tmax | 0-72h
t1/2 | 0-72h
AUCinf | 0-72h

CONTACTS AND LOCATIONS:
Overall Officials: JaeWook Ko, M.D., Principal Investigator — Samsung Seoul Hospital
Locations (1):
- Samgsung Seoul Hospital, Seoul, South Korea